CLINICAL TRIAL: NCT06616155
Title: Study of JAK Inhibition in Stem-Like Prostate Cancer (JASPER): A Phase 1b/2a Multicenter Study of Ruxolitinib and Enzalutamide in Castration Resistant Prostate Cancer
Brief Title: Ruxolitinib and Enzalutamide for the Treatment of Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2023.109; NCI-2024-06533 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00249478
Record Dates: First submitted 2024-08-31; First posted 2024-09-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Specimen Handling; enzalutamide; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ruxolitinib, enzalutamide) (Experimental): Patients receive ruxolitinib PO BID and enzalutamide PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, CT and bone scan throughout the study. Patients may also undergo a tissue biopsy on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Enzalutamide; Drug: Ruxolitinib

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV 3100; MDV-3100; MDV3100; Xtandi
Drug: Ruxolitinib — Given PO
  Other Names: INCB 018424; INCB-018424; INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424

SUMMARY:
This phase I/II tests the safety, side effects and best dose of ruxolitinib in combination with enzalutamide and how well it works in treating patients with prostate cancer that remains despite blocking hormone production (castration-resistant) and that has spread from where it first started to other places in the body (metastatic). Ruxolitinib, a kinase inhibitor, slows down the growth of the tumor by blocking the proteins, JAK1 and JAK2, tumors use to grow. Enzalutamide, an androgen receptor inhibitor, works by blocking the effects of androgen (a male reproductive hormone). This may help stop the growth and spread of tumor cells that need testosterone to grow. Giving ruxolitinib in combination with enzalutamide may be safe, tolerable, and/or effective in treating metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information prior to registration
* Males age ≥ 18 years with progressive metastatic, castration-resistant prostate cancer, previous adenocarcinoma histology confirmation required
* Ability to understand a written informed consent document, as determined by the study physician or designee
* Surgical castration or continuous medical castration ≥ 8 weeks prior to screening; serum testosterone < 50 ng/dL
* Have progressed on prior abiraterone treatment by Prostate Cancer Working Group 3 prostate specific antigen (PSA) criteria

  * PSA must rise on two measurements at least 1 week apart in order to be eligible. Refer to PCWG3 for clarification.
  * Most Recent absolute PSA must be > 2.0 ng/mL
* Patient meets definition of poor responder to abiraterone by one of the following:

  * Abiraterone started in hormone-sensitive prostate cancer (HSPC) disease setting (abiraterone started within 4 months of starting continuous androgen deprivation therapy [ADT]): < 12 months duration on abiraterone
  * Abiraterone started in castration-resistant prostate cancer (CRPC) disease setting: < 6 months duration on abiraterone due to progression or failure to achieve PSA50 response while on therapy
* The patient's current or most recent treatment is ADT and abiraterone. Participants must sign consent within 30 days of discontinuing abiraterone or prior to stopping abiraterone
* Patients must be willing to undergo metastatic tumor biopsy during screening. If no metastatic lesion is safely accessible to tumor biopsy, this requirement will not be required
* 50% of patients must have measurable disease by RECIST 1.1 criteria

  * Once 50% of total expected cohort has non-measurable disease, only patients with measurable disease by RECIST 1.1 criteria will be eligible. (Percentages with measurable disease are not relevant within dose escalation. Once dose expansion is started, those at expansion dose would be included in percentage evaluation.)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2 (grade 2 ECOGs should be related to disease and thus potentially reversible)
* A male participant must agree to use of contraception during the treatment period and for at least 90 days after the last dose of study drug. Female partners of male patients should also use contraception for 90 days after the last dose of study drug if they are of childbearing potential
* Platelets ≥ 125,000/mm^3 (obtained within 28 days prior to starting study therapy) (if creatinine clearance [CrCl] is between 30-59, the platelet entry criteria is > 150,000/mm^3)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained within 28 days prior to starting study therapy)
* Hemoglobin ≥ 11 g/dL (obtained within 28 days prior to starting study therapy) No transfusions within 90 days prior to screening unless performed for acute bleeding
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN) (obtained within 28 days prior to starting study therapy) For patients with known liver metastasis: (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN
* Bilirubin ≤ 1.5 the upper limit of normal (ULN) OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 x ULN. For subjects with known Gilbert's disease, bilirubin ≤ 3.0 mg/dL (obtained within 28 days prior to starting study therapy)
* Creatinine clearance (CrCl) ≥ 30 mL/min (obtained within 28 days prior to starting study therapy) For creatinine clearance estimation, the Cockcroft and Gault equation should be used

Exclusion Criteria:

* History of untreated (with radiotherapy and/or surgery) brain metastasis is not allowed (stable and treated metastases are allowed)
* History of seizures or known hypersensitivity to enzalutamide, ruxolotinib or any of the excipients in the product
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with the absorption of the study medications
* Uncontrolled hypertension as indicated by systolic blood pressure (SBP) > 170 mmHg or diastolic blood pressure (DBP) > 105 mmHg on 2 consecutive measurements at screening visit unless known to have white coat hypertension syndrome
* Have received chemotherapy in the metastatic castration-resistant setting (docetaxel within the hormone sensitive setting is allowed)
* Failure to recover to grade 1 or lower toxicity related to prior systemic therapy (excluding alopecia and neuropathy) prior to study consent
* Current active infection with any of the following: hepatitis B, hepatitis C, active tuberculosis, latent tuberculosis. Patients with well controlled HIV are eligible however all drug interactions with HIV drug and study therapies have to be reviewed
* History of myocardial infarction, stroke, pulmonary embolism or deep vein thrombosis within 6 months of study enrollment
* Study physician estimates life expectancy less than 6 months or patient is unable to swallow medications
* Patients currently taking fluconazole
* Currently receiving supplements containing androgens or medications known to be strong inhibitors of CYP2C8, strong inducers (except enzalutamide) or strong inhibitors of CYP3A4 and substrates of CYP3A4, CYP2C9 and CYP2C19 with a narrow therapeutic window. If substitution is possible, strong inducers, inhibitors and substrates must be discontinued at least 7 days or 5 half-lives (which ever longer) prior to the first administration of enzalutamide
* Due to risk of tuberculosis (TB) reactivation, patients deemed at high risk by treating provider (e.g., close contact with someone with active TB, history of active/latent TB) should be excluded
* Those with underlying hepatic disease with a CHILD-PUGH class A, B or C impairment are excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days
  DLT will be defined based on the rate of drug-related grade 3-5 adverse events (AEs) experienced. AEs will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The proportion of patients at each dose level experiencing each grade level of toxicity will be described. To estimate the frequency and severity of AEs associated with treatment, the proportion of subjects encountering toxicity at each dose level will be reported with exact 95% binomial confidence intervals.
Maximum tolerated dose (MTD) | Up to 28 days
  MTD will be defined based on the rate of drug-related grade 3-5 adverse events (AEs) experienced. MTD will be the highest dose level at which the probability of a subject experiencing a DLT during cycle 1 falls between 0.23 and 0.33.

SECONDARY OUTCOMES:
Prostate specific antigen (PSA) reduction of 50% (PSA50) rate | Up to 6 months
  PSA50 response will be defined by at least 50% decline in PSA level from baseline measured at least 3 weeks apart.
Objective response rate (ORR) | Up to 6 months
  ORR will be defined as the proportion of subjects who experience radiographic response (complete response or partial response by Response Evaluation Criteria in Solid Tumors 1.1 criteria). Proportion of participants with ORR will be estimated along with corresponding 2-sided exact 95% Clopper-Pearson.
Incidence of AEs | Up to 30 days after last dose of study treatment
  AEs will be assessed and graded according to CTCAE version 5.0. To estimate the frequency and severity of AEs associated with treatment, the proportion of subjects encountering toxicity at each dose level will be reported with exact 95% binomial confidence intervals.
Objective progression free survival (PFS) | At start of treatment until clinical progression, death or radiographic progression, assessed up to 2 years
  PFS will be defined by Prostate Cancer Working Group 3 criteria. Median PFS will be estimated by the Kaplan-Meier method and corresponding 95% confidence interval will be derived.

OTHER OUTCOMES:
Pharmacokinetics (PK) Cmax | Up to 30 days after last dose of study treatment
  PK will be assessed via measurement in plasma at pre-specified timepoints. PK analysis will be performed on individual serum concentration data. Serum concentrations will be listed and summarized using descriptive statistics.
Phosphorylated STAT3 (pSTAT3) percentage | Up to 30 days after last dose of study treatment
  Pharmacodynamics will be assessed through measurement of pSTAT3 percentage in whole blood at pre-specified timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Zachery R Reichert, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (3):
- United States (3):
  - Rush University, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No